CLINICAL TRIAL: NCT03595202
Title: Phase I Clinical Study of TS-143 in Healthy Adult Male Subjects (Multiple-Dose Administration)
Brief Title: Clinical Study of TS-143 in Healthy Adult Male Subjects (Multiple-Dose Administration)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TS143-01-03
Record Dates: First submitted 2018-04-18; First posted 2018-07-23 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2018-07

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Step1:4㎎ TID (Other): TS-143 12mg total dose/day or Placebo
  Interventions: Drug: TS-143; Drug: Placebo
- Step2:11㎎ TID (Other): TS-143 33mg total dose/day or Placebo
  Interventions: Drug: TS-143; Drug: Placebo

INTERVENTIONS:
Drug: TS-143 — Subjects should take 4 capsules once and 3 times per day in step 1. Subjects should take 2 capsules once and 3 times per day in step 2.
Drug: Placebo — Subjects should take 4 capsules once and 3 times per day in step 1. Subjects should take 2 capsules once and 3 times per day in step 2.

SUMMARY:
To investigate the safety, pharmacokinetics and pharmacodynamics of TS-143 when administered 3 times a day for 10 days to healthy Japanese adult males using placebo-controlled, double-blind, dose escalation study design.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a BMI of 18.5 to less than 25.0 at the time of the screening tests
* Subjects judged by the principal investigator or a subinvestigator to be appropriate for participation in the study based on the results of the screening tests and the tests conducted before the investigational drug treatment on Day 1
* Subjects capable of receiving an explanation of this study before participation, understanding the details, and providing written informed consent themselves

Exclusion Criteria:

1. Subjects meeting any of the following criteria in the results of screening tests, tests conducted on the day before the first investigational treatment (Day -1), and tests conducted before the investigational drug treatment on the morning of Day 1:

   * Red blood cell count: ≥535 × 10^4 /μL
   * Hemoglobin: ≥16.2 g/dL
   * Hematocrit: ≥47.5%
   * Reticulocyte rate: Outside of the reference value range
2. Subjects meeting any of the following criteria in the screening tests:

   * Serum EPO concentration: Outside of the reference value range
   * Ferritin: ≤30 ng/mL or >upper limit of the reference value
3. Subjects meeting any of the following criteria in the vital signs in the screening tests and the tests conducted before the investigational drug treatment on the morning of Day 1:

   * Blood pressure: Systolic blood pressure ≥140 mmHg, or diastolic blood pressure ≥90 mmHg
   * Pulse rate: <40 bpm, or ≥100 bpm
   * Body temperature: ≥37.5°C

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Incidence of subjects with adverse events | 18 days
  To evaluate the safety of TS-143 given single administration in healthy volunteers by incidence of subjects with adverse events which include abnormal electrocardiograms, vital signs, and clinical laboratory parameters.
Plasma concentrations of unchanged form (ng/mL) | 13 days
Urinary excretions of unchanged form (ng/mL) | 12 days
Serum EPO concentration | 13 days
Reticulocyte count | 13 days
Plasma vascular endothelial growth factor (VEGF) concentration | 13 days
Serum iron (μg／dL) | 13 days
Total iron binding capacity（μg／dL） | 13 days

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Okuyama, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No